CLINICAL TRIAL: NCT04234620
Title: A Prospective, Single-arm, Multicenter, Non-interventional Real-world Study of Toripalimab Injection in the Treatment of Malignant Tumors in Chinese Population.
Brief Title: Intensive Medicines Monitoring Study of Toripalimab Monoclonal Injection (Tuoyi) .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: JS001-PMS-CO1
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Melanoma; Lung Cance; Breast Cancer
MeSH Terms: conditions — Melanoma; Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Toripalimab injection: Use of Toripalimab injection in the real world
  Interventions: Drug: Toripalimab injection

INTERVENTIONS:
Drug: Toripalimab injection — 240 mg/6 mL/vial. The recommended dose of Toripalima is 3 mg/kg, intravenous infusion every 2 weeks until disease progression or intolerable toxicity.

SUMMARY:
This study was a prospective, single-arm, multi-channel, multicenter, non-interventional real-world study to evaluate the safety and efficacy of Toripalimab injection in the treatment of unresectable or metastatic melanoma with previously systemic failure . The study population currently included only in the melanoma cohort-unresectable or metastatic melanoma patients who had previously failed systemic therapy. If new indications are approved during the implementation of the project, patients with new indications using Toripalimab injection will also be included in this study as a new cohort.This study uses offline (physical hospital) and online (DTP pharmacy and Lingke (Yinchuan) Internet hospital) to collect data and information, relying on Lingke technology (Beijing) Co., Ltd. EDC (Medical Research Cloud) database for data collection and processing. The classification of adverse events was based on the general toxicity evaluation standard NCI CTCAE 5.0 of the National Institute of Oncology (Chinese version).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with approved indications of Toripalimab injection;
2. Patients treated with Toripalimab injection;
3. Patients who agreed to participate in this study and signed an informed consent form.

Exclusion Criteria:

1. Refused to participate or refused to cooperate with the procedure;
2. Those who participated in the intervention study of other unapproved drugs / therapies and less than 5 half-lives after the last use of the study drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population currently included only in the melanoma cohort-unresectable or metastatic melanoma patients who had previously failed systemic therapy. If new indications are approved during the implementation of the project, patients with new indications using Toripalimab injection will also be included in this study as a new cohort.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-07-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of all ADR. | 3 years
  the incidence of all ADR: the number and percentage of patients with ADR, and the number of ADR events will be summarized according to the International Medical Dictionary (MedDRA) preferred terminology and adverse events General terminology Standard (NCI CTCAE5.0 Chinese version). Any ADR collected during the study will be included in the ADR summary.
known ADR. | 3 years
  The incidence of known adverse reactions ((ADR)).
The occurrence of new adverse reactions ((ADR) | 3 years
  The occurrence of new adverse reactions ((ADR)).
SADR | 3 years
  The incidence, severity and risk factors of severe adverse reactions ((SADR)).
Immune-related ADR | 3 years
  The incidence, severity and risk factors of immune-related adverse reactions.
The incidence of adverse drug reactions ((ADR)) in special populations. | 3 years

SECONDARY OUTCOMES:
AE | 3 years
  1. the incidence of all adverse events (AE);
  2. the incidence of different severity AE;
SAE | 3 years
  The incidence of severe adverse events (SAE):
Immune-related AE. | 3 years
  The incidence, severity of immune-related adverse events;
1 -, 2 -, 3-year OS rate. | 3 years
  Survival indicators: overall survival (OS); 1 -, 2 -, 3-year OS rate.

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - The first affiliated Hospital of Jinlin Universtiy, Changchun
  - Hunan cancer hospital, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Chongqing Haijiya Cancer Hospital, Chongqing
  - Fujian province cancer hospital, Fuzhou
  - Zhejiang cancer hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Qilu Hospital of Shandong university, Jinan
  - Shandong province cancer hospital, Jinan
  - Affiliated Cancer Hospital of Guangxi Medical university, Nanjing
  - Najing Drum Tower Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanxi Bethune Hopital, Shanxi
  - The fouth Hospital of Hebei Medical University, Shijiazhuang
  - The Second affiliated Hospital of Suzhou Universtiy, Suzhou
  - Tianjin Medical University cancer institute & Hospital, Tianjin
  - Hubei cancer hospital, Wuhan
  - Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - Wuhan Union Hospital, Wuhan
  - The first affiliated Hospital of Xiamen Universtiy, Xiamen
  - Yinchuan Lingke Internet Hosipital, Yinchuan
  - Affiliated Hopital of Guangdong Medical University, Zhanjiang
  - Henan cancer hospital, Zhengzhou